CLINICAL TRIAL: NCT04877158
Title: Pilot Intervention for Attribution Biases in Eating Disorders
Brief Title: Pilot Intervention for Social Biases in Eating Disorders
Acronym: SBPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Carrie McAdams, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-042016-079
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Intervention Model Description: Self-concept measures (Attribution Biases, Self-Esteem) and psychological symptoms (Eating, depression, anxiety) will be assessed before and after completion of the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-Blame and Perspective-Taking Intervention (Experimental): These participants are enrolled with intent to participate in the group therapy intervention.
  Interventions: Behavioral: Self-Blame and Perspective-Taking Intervention

INTERVENTIONS:
Behavioral: Self-Blame and Perspective-Taking Intervention — The intervention is a group therapy that consists of experiential art tasks followed by psychoeducation about social behaviors with weekly homework. There are four sessions, each one week apart.

SUMMARY:
Both behavioral, psychological, and cognitive differences related to social cognitive function have been related to illness-state in eating disorders, but interventions that directly target these problems are limited. This pilot intervention explores whether a brief art-therapy team-building intervention coupled with psychoeducation about social behavior can change self-concept or clinical symptoms in patients with eating disorders. Participants will complete pre-treatment assessments related to social behaviors and clinical symptoms, attend four two-hour group sessions, and provide two follow-up post-treatment assessments at 1-4 weeks after the treatment and 3-5 months later. Comparisons between the pre-intervention data and the first follow-up will be the primary outcome measures. The primary hypotheses are that participants will show increases in self-esteem and positive self-attributions and decreases in eating disorder symptoms after the intervention. The secondary hypothesis is that other clinical symptoms (depression, anxiety) will be improved after the intervention. Feedback from participants about their experience with the study will assess perceived benefits as well as acquisition of the psychoeducation targets.

DETAILED DESCRIPTION:
This project will recruit subjects with eating disorders in the Dallas Fort Worth area. Pre-assessment measures of anxiety, self-esteem, depression, eating disorder symptoms, and attributional style will be completed before the intervention. Participants attend four weekly sessions of a group psychoeducational intervention. The intervention includes an art therapy experiential activity, psychoeducation on social function, reflection and discussion of sample videos and scripts, homework assignments, and guided discussions. Post-assessments will be completed 1-4 weeks and 3-5 months after the interventions is completed.

A. Intake and Screen: Screening checklist for ED symptoms. Demographic Sheet; Clinical History (low BMI); Mini-International Neuropsychiatric Interview for DSM-V (MINI); Eating Disorder Assessment for DSM-V (EDA-5); Wechsler Abbreviated Scale of Intelligence (WASI)

B. Pre/Post Measures (Done at three time points, Pre:1-4 weeks before intervention; Post1: 1-4 weeks after intervention; and Post2: 3-5 months after intervention).

1. Internal, Personal, and Situational Attribution Questionnaire, (IPSAQ)
2. State Self-Esteem Scale (SSE)
3. Trait Self-Esteem Scale (TSE)
4. Eating Disorder Examination Questionnaire, (EDE-Q)
5. The Quick Inventory of Depression, Clinician-Rated (QIDS)
6. Structured Interview Guide for Hamilton Anxiety Scale (SIGH-A)

C. Feedback about the intervention is obtained from queries immediately after the last session and at the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* eating disorder, current or recent
* female
* appropriate for partial hospital, intensive outpatient or outpatient treatment

Exclusion Criteria:

* medically unstable
* in inpatient or residential treatment

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants only
Enrollment: 29 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Change in self- attribution (externalizing bias score) from Pre-assessment to Post-assessment 1 | Baseline, 4 weeks after intervention
  Internal Personal Situational Attributions Questionnaire (IPSAQ) measures externalizing bias (EB) that is calculated by subtracting the number of internal attributions for negative events from the number of internal attributions for positive events. A positive EB score indicates strong self-serving bias (blaming oneself less for negative events than for positive events).
Change in state self-esteem score from Pre-assessment to Post-assessment 1 | Baseline, 4 weeks after intervention
  State Self-Esteem Scale measures a participant's self-esteem at a given point in time. Possible scores range from 0-5 with higher scores indicating better outcome.
Change in trait self-esteem score from Pre-assessment to Post-assessment 1 | Baseline, 4 weeks after intervention
  Rosenberg trait self-esteem scale measures trait self-esteem (TSE). Possible scores range from 0-4 (from 1: strongly disagree, to 4: strongly agree), with higher scores indicating higher TSE.
Study components feedback score | 4 weeks after starting intervention
  The Attribution Bias Intervention Questionnaire addressed study component feedback using both a rating scales and free form written commentary. Possible scores range from 1 to 10 with higher scores indicating more positive values.
Patient satisfaction score | 5-9 weeks after intervention
  The Attribution Bias Feedback Form measured patient satisfaction (the impact and value of study) with free-form verbal responses as well as a single rating scale. Possible scores range from 1 to 5 with higher scores indicating more satisfaction with the intervention.
Change in eating disorder symptoms score from Pre- assessment to Post-assessment 1 | Baseline, 4 weeks after intervention
  The Eating Disorder Examination Questionnaire measures the severity of eating disorder symptoms. Possible scores on global eating disorder pathology range from 0 to 6 with higher scores indicating more severity of eating disorder, with scores of 2 or less typical of normative eating behavior/cognitions and scores of 2 to 6 are consistent with eating disorder symptoms, with higher scores suggesting more types of disordered eating are present.

SECONDARY OUTCOMES:
Change in depression symptoms scores from Pre-assessment to Post-assessment 1 | Baseline, 4 weeks after intervention
  QIDS (Quick Inventory of Depressive Symptoms) measures depression symptoms. Possible scores range from 0-27, with scores of 5 or lower indicative of no depression, scores from 6 to 10 indicating mild depression, 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression.
Change in depression symptoms scores from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention
  QIDS (Quick Inventory of Depressive Symptoms) measures depression symptoms. Possible scores range from 0-27, with scores of 5 or lower indicative of no depression, scores from 6 to 10 indicating mild depression, 11 to 15 indicating moderate depression, 16 to 20 reflecting severe depression, and total scores greater than 21 indicating very severe depression.
Change in anxiety symptoms score from Pre-assessment to Post-assessment 1 | Baseline, 4 weeks after intervention
  SIGH-A (Structured Clinical Interview for Hamilton Anxiety Scale) measures Anxiety symptoms. Possible scores range from 0-56 with score of 0 means no anxiety symptom. ( <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Lower scores indicate better outcome)
Change in anxiety symptoms score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention
  SIGH-A (Structured Clinical Interview for Hamilton Anxiety Scale) measures anxiety symptoms. Possible scores range from 0-56 with score of 0 means no anxiety symptom ; <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Lower scores indicate better outcome.
Change in eating disorder symptoms score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention
  The Eating Disorder Examination Questionnaire measures the severity of eating disorder symptoms. Possible scores on global eating disorder pathology range from 0 to 6 with higher scores indicating more severity of eating disorder, with scores of 2 or less typical of normative eating behavior/cognitions and scores of 2 to 6 are consistent with eating disorder symptoms, with higher scores suggesting more types of disordered eating are present.
Change in self- attribution (externalizing bias score) from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention
  Internal Personal Situational Attributions Questionnaire (IPSAQ) measures externalizing bias (EB) that is calculated by subtracting the number of internal attributions for negative events from the number of internal attributions for positive events. A positive EB score therefore indicates strong self-serving bias (blaming oneself less for negative events than for positive events).
Change in state self-esteem score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention
  State self-esteem scale measures a participant's self-esteem at a given point in time. Possible scores range from 0-5 with higher scores indicating better outcome.
Change in trait self-esteem score from Pre-assessment to Post-assessment 2 | Baseline, 3-5 months after intervention
  Rosenberg trait self-esteem scale measures Trait Self-Esteem (TSE). Possible scores range from 0-4 (from 1: strongly disagree, to 4: strongly agree), with higher scores indicating higher TSE.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie McAdams, MD PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UTSW, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hagan WS, Mericle S, Hunt BJ, Harper JA, Palka JM, Pelfrey S, McAdams CJ. Qualitative patient experiences from the Self-Blame and Perspective-Taking Intervention for eating disorders. J Eat Disord. 2021 Oct 14;9(1):127. doi: 10.1186/s40337-021-00483-9. PMID 34649621